CLINICAL TRIAL: NCT06241521
Title: Myasthenia Gravis Registry in China
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: China Alliance for Rare Diseases (Unknown); National Center for Neurological Disorders (China) (Unknown); China myasthenia gravis collaborating group (CMGCG) (Unknown)
Responsible Party: Principal Investigator, Chongbo Zhao, Vice President, Huashan Hospital
Other Study IDs: 2023M-022; 2022YFC3501303 (Other Grant/Funding Number: China's National Key R&D Program); 82071410 (Other Grant/Funding Number: National Natural Science Foundation of China); 82001335 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Prospective study; Observational study; Patient registry
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood, Plasma, Serum, Blood RNA extraction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myasthenia gravis patients

SUMMARY:
Myasthenia gravis (MG) is an autoimmune disease caused by dysfunction at the neuromuscular junction, characterized by partial or generalized skeletal muscle weakness and fatigability. The estimated annual incidence rate of MG in China is 0.68/100,000, with a high rate of relapse and poor treatment compliance. This study is a prospective, observational, multi-center patient registry across China. To support standardized management and follow-up of MG patients in China, a Cloud-based MG Patient Management Platform (CN MG Base) was established in September 2023 with the support of the Chinese Rare Diseases Alliance. The platform aims to collect longitudinal clinical data including demographic information, age of onset, medical history, comorbidities, medication usage, treatment responses, and others. It is intended to collect newly registered MG cases each year and follow up with these patients at one-year intervals for ten years

DETAILED DESCRIPTION:
This study is a observational nationwide multicenter MG registry research. Starting from the baseline, annual follow-ups will be conducted to prospectively collect information on treatment medications, prognosis, and safety events. The following classification definitions can be applied: ① MG clinical subtypes (ocular, early-onset generalized, thymoma-related, late-onset generalized, MuSK-related, and seronegative); ② Different treatment methods (classic immunotherapy group, B-cell-targeted therapy, complement inhibition therapy, rapid-acting therapy, and IL-6 pathway inhibitors, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Fluctuating weakness in skeletal muscles, such as extraocular, bulbar, limb muscles, etc.. Demonstrating fluctuation and fatigability: Weakness is usually worse in the morning and improves with rest; worsens with sustained activity.
* Patients themselves or their guardians can understand and sign the informed consent form.

To meet the eligibility criteria, at least one of the following additional criteria must be met:

* a. Positive Tensilon test;
* b. Decrease in compound muscle action potential by more than 10% with low-frequency repetitive nerve stimulation or widening of the "jitter" (the variability in time of the second action potential relative to the first) on single-fiber electromyography, with or without blocking;
* c. Positive antibodies: Serum testing positive for AChR antibodies, MuSK antibodies, or LRP4 antibodies.

Exclusion Criteria:

* Patients with mental illness who cannot cooperate.
* Patients with multiple organ dysfunction or in extremely critical condition, unable to complete relevant medical history collection or evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MG patients mostly of Chinese Han ethnicity (ocular MG type no more than 30%).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2034-02-01 (Estimated); Study Completion 2035-01-30 (Estimated)

PRIMARY OUTCOMES:
MSE proportion | Ten years
  The proportion of patients achieving minimal symptom expression (MSE, defined as reaching an ADL score of 0 or 1) after treatment.

SECONDARY OUTCOMES:
Safety events | Ten years
  Safety events including upper respiratory tract infection, lower respiratory tract infection, urinary tract infection, and other infections;
Relapse of MG symptoms | Ten years
  Having reached MSE for over a year but experiencing a symptom relapse, manifested as an increase in ADL score greater than or equal to 2 points.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Xuanwu hospital, Capital medical university, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya hospital, Central south university, Changsha, Hunan
  - The First Hospital, Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital, Jilin University, Changchun, Jilin
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tangdu Hospital, The Air Force Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality